CLINICAL TRIAL: NCT06090188
Title: Feasibility of a Culture-Based Multicomponent Cognitive Training Program in Older People With Dementia: A Randomized Controlled Pilot Study
Brief Title: Culture-Based Multicomponent Cognitive Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Su-Hsien Chang, Professor, National Tainan Junior College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NTJCN 1121003
Record Dates: First submitted 2023-10-04; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Nursing Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Subjects in the experimental group received a series of culture-based multicomponent cognitive training activities via research assistants (RAs) and caregivers of the centres for 8 weeks, then provided by caregivers of the day care centre for 8 weeks with RAs providing assistance with the activity process.
  Interventions: Other: A Culture-Based Multicomponent Cognitive Training Program
- comparison group (Active Comparator): Participants in the comparison group received these activities via two RAs and day care caregivers for 16 weeks.
  Interventions: Other: A Culture-Based Multicomponent Cognitive Training Program

INTERVENTIONS:
Other: A Culture-Based Multicomponent Cognitive Training Program — Activities of the program were structured, cognitive, leisure activities based on Chinese and Taiwanese culture for cognitively impaired older people. Activities contained structured brain-exercise activities and musical activities. The structured brain-exercise activities included playing musical instruments or singing, playing board games, and classes in Chinese, sciences, sociology, physical education, cooking, and math. Chinese and Taiwanese cultures were included within the structured brain-exercise activities curriculum, such as food, clothing, architecture, places of interest, folklore, etiquette, celebrations, religion, art, etc. Participants began with a musical exercise, then had 20-30 minutes of physical exercise with 5 minutes of warm-up at the beginning and 5 minutes of cool down. The program was provided for at least 40-60 minutes, twice a week, for 8 weeks via RAs and day centre caregivers.

SUMMARY:
To provide care without exacerbating behavioral and psychological problems and preventing functional decline, a multi-component, cognitive training program was designed. The purpose of this study is to test the effectiveness of this multi-component, cognitive training program in day care centers for elderly people with dementia to prevent cognitive function decline, self-care abilities decline, and behavior problems or the development of depressive moods.

DETAILED DESCRIPTION:
The purpose of the study is to test the effectiveness of this multi-component, cognitive training program in day care centers for elderly people with dementia to prevent cognitive function decline, self-care abilities decline, and behavior problems or the development of depressive moods. This study was a 4-month cluster-randomized controlled trail. Participants who met sample selection criteria were recruited and assigned to either the experimental group or the comparison group, depending on the day-care center they attended. Subjects in the experimental group were received with the multi-component, cognitive training program (MCCTP) via research assistants (RAs) and caregivers of day care center for 8 weeks, then provide by caregivers of day care center for 8 weeks, as well as RAs provided assistance for activity process.

ELIGIBILITY:
Inclusion Criteria:

1. persons aged 60 years and over, (2) living in their own home, (3) with or without a hearing device and able to speak Mandarin or Taiwanese, (4) attending a day care centre at least three days per week, (5) cognitively impaired as determined by a score of 22 or lower on the Mini-Mental State Examination (MMSE), and (6) self or legal proxy agreed to participate in the study.

Exclusion Criteria:

- Persons were excluded if they were bedridden and unable to sit in a wheelchair or had one or more acute illnesses during the data collection period causing them to be unable to return to the day care centre.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function | baseline, 8 weeks post-intervention, 16 weeks post-intervention
  The Mini-Mental State Examination (MMSE) was used to measure the cognitive status of the participants. It was collected through individual interviews. The MMSE is a criterion-referenced instrument that contains 11 items. It can be used to examine a person's orientation, registration, recall, attention, calculation ability, understanding and use of language, and praxis. The score ranges from 0 to 30. The sum of the score is used to stratify cognitive function (Crun, Anthony, Bassett, & Folstein, 1993).
Behavioural problems | baseline, 8 weeks post-intervention, 16 weeks post-intervention
  The Clifton Assessment Procedures for the Elderly - Behaviour Rating Scale (CAPE-BRS) was used to measure behavioural problems, including activities of daily living, apathy, communication difficulties, and social disturbance. It was collected by observations. The CAPE-BRS includes 18 items; each item is scored from 0 to 2. The total score ranges from 0 to 36. Higher scores indicate greater disability (Pattiem & Gilleard, 1979).
Symptoms of depression | baseline, 8 weeks post-intervention, 16 weeks post-intervention
  The Cornell Scale for Depression in Dementia (CSDD) was used to examine symptoms of depression. It was collected by observations. It includes 19 items and measures mood-related signs, behavioural disturbances, physical signs, cyclic functioning, and ideational disturbance. The total score ranges from 0 to 38. A score from 0 to 6 indicates no depression, 7 to 9 indicates mild depression, 10 to 19 indicates possible severe depression, and 18 and over indicates severe depression. The CSDD has been translated into Chinese, and the validity and reliability have been examined (Sharp & Lipsky, 2002).
Self-care abilities | baseline, 8 weeks post-intervention, 16 weeks post-intervention
  The Refined ADL Assessment Scale (RADL) was used in this study to measure the performance of activities of daily living (ADLs). It was collected by observations. The RADL is designed to measure 5 tasks of basic ADLs for older adults with Alzheimer's and related disorders. It includes tasks of feeding, washing, grooming, dressing, and toileting. The toileting task was not assessed in this study because it was likely to disturb the privacy of older adults. Each task in the RADL is broken down into 2 to 5 subtasks. Each subtask is further broken down into the sequence of steps needed for the completion of the activity. The scores for the feeding activity range from 0 to 126, for the washing activity range from 0 to 204, for the grooming activity range from 0 to 174, and for the dressing activity range from 0 to 150. A higher score indicates greater independence in ADL performance.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Ah Lian Day Care Center, Kaohsiung City
  - Anping Day Care Center, Tainan
  - Huishan community long-term care institution, Tainan
  - Meiyu East District Day Care Center, Tainan

IPD SHARING:
Plan to Share IPD: No